CLINICAL TRIAL: NCT03617575
Title: The Effect of Apo- and Holo-Lactoferrin and Dosing Regimen on Iron Absorption From a Maize-based Porridge in Kenyan Infants
Brief Title: The Effect of Lactoferrin and Dosing Regimen on Iron Absorption From a Maize-based Porridge in Kenyan Infants
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Swiss Federal Institute of Technology (Other)
Responsible Party: Principal Investigator, Prof. Michael B. Zimmermann, Head of Laboratory of Human Nutrition, Swiss Federal Institute of Technology
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: Fe_LF
Record Dates: First submitted 2018-07-24; First posted 2018-08-06 (Actual); Last update posted 2020-05-13 (Actual); Status verified 2020-05

CONDITIONS: Iron-deficiency
MeSH Terms: conditions — Anemia, Iron-Deficiency | interventions — hololactoferrin, human

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- apo-Lactoferrin (Placebo Comparator): unsaturated (= no iron) form of Lactoferrin Lactoferrin is a bovine milk protein Test Meal A1
  Interventions: Dietary Supplement: apo-Lactoferrin
- holo-Lactoferrin (Placebo Comparator): saturated (= contains a certain amount of iron) form of Lactoferrin Lactoferrin is a bovine milk protein Test Meal B1
  Interventions: Dietary Supplement: holo-Lactoferrin
- FeSO4 (Placebo Comparator): Ferrous sulfate = FeSO4 acting as the reference Test Meal C1
  Interventions: Dietary Supplement: FeSO4
- 1. FeSO4 (Placebo Comparator): Ferrous sulfate = FeSO4 Test Meal A2
  Interventions: Dietary Supplement: 1. FeSO4
- FeSO4 after 1 day break (Placebo Comparator): Ferrous sulfate = FeSO4 Test Meal B2
  Interventions: Dietary Supplement: FeSO4 after 1 day break
- FeSO4 after 2 day break (Placebo Comparator): Ferrous sulfate = FeSO4 Test Meal C2
  Interventions: Dietary Supplement: FeSO4 after 2 day break

INTERVENTIONS:
Dietary Supplement: apo-Lactoferrin — 1.41 g of apo-Lactoferrin will be given together with 1.42 mg FeSO4 (0.08 mg of iron naturally in apo-Lf [total of 1.5 mg iron]) in a maize porridge (extrinsically labeled)
  Arms: apo-Lactoferrin
Dietary Supplement: holo-Lactoferrin — 1.41 g of holo-Lactoferrin (intrinsically labeled with 1.5 mg 57Fe) will be given together in a maize porridge
  Arms: holo-Lactoferrin
Dietary Supplement: FeSO4 — 1.5 mg FeSO4 as 54Fe in a maize porridge
  Arms: FeSO4
Dietary Supplement: 1. FeSO4 — 10 mg 56Fe + 2 mg 54Fe Is the 1. FeSO4 meal in maize porridge
  Arms: 1. FeSO4
Dietary Supplement: FeSO4 after 1 day break — 10 mg 56Fe + 2 mg 57Fe Is the 2. FeSO4 in maize porridge with a 1 day washout period
  Arms: FeSO4 after 1 day break
Dietary Supplement: FeSO4 after 2 day break — 10 mg 56Fe + 2 mg 58Fe Is the 3. FeSO4 in maize porridge with a 2 day washout period
  Arms: FeSO4 after 2 day break

SUMMARY:
The purpose of this study is to measure iron absorption from maize-based porridge fortified with either apo-lactoferrin, holo-lactoferrin or ferrous sulfate and to test whether there is an effect of these. Additionally, iron absorption from maize-based porridge containing 12 mg ferrous sulfate will be measured when consumed every other day versus every third day.

DETAILED DESCRIPTION:
Infants and young children in sub-Saharan Africa have high rates of iron deficiency anemia (IDA), which adversely affects their growth and cognitive development. In-home iron fortification of complementary foods using micronutrient powders (MNPs) reduces risk for IDA by ensuring that the iron needs of infants and young children are met without changing their traditional diet. Oral iron syrups, typically containing iron as ferrous sulfate, can also be given to prevent/correct IDA. However, iron absorption from MNPs and iron syrups, particularly when given with complementary foods high in inhibitors of iron absorption, is low. Thus, there is a need to find iron formulations with higher bioavailability for use in African infants. In a recent trial in Kenya, the investigators demonstrated that a prebiotic could improve iron bioavailability from an iron-containing MNP.

In this study, the investigators plan to assess the human milk compound lactoferrin (Lf) as a possible enhancer of iron absorption. Lf is an important iron-binding protein in human milk, which has been thought to be responsible for the high bioavailability of breast-milk iron. It has many biological functions, including iron absorption, antimicrobial activity, immunomodulatory effects and stimulatory effect on cell proliferation. Lf has different iron binding statuses: the iron free form (apo-Lf) and the iron-saturated form (holo-Lf). One of the two main biological activities of Lf provided by the diet is the control of iron uptake, which is mediated by the Lf receptor (LFR) as undigested Lf can bind to LFR and facilitate the uptake of iron. Therefore, Lf may be a nutritional iron source and may enhance iron absorption in infants. To evaluate the possible role of Lf on the availability of iron, iron absorption will be measured from bovine Lf (bLf). BLf has GRAS (generally considered as safe) status by the US Food and Drug Administration.

To optimize iron absorption, timing of supplementation might as well be important. Hepcidin, a key regulator of systemic iron balance and a single dose of iron can increase hepcidin levels and potentially inhibit iron absorption from a second dose, consumed close in time to the first dose. The investigators will conduct two studies, where 24 infants aged 3-14 months in Msambweni, Kenya, will be enrolled. In study 1, on three alternate mornings, these infants will consume maize porridge containing a low iron dose (1.5 mg) to compare iron absorption between meals with apo-Lf, holo-Lf and ferrous sulfate (FeSO4) as a reference; and whether the addition of either apo- or holo-Lf has a beneficial effect on iron absorption. The investigators hypothesize that iron absorption will be higher when holo-Lf is present in the meal compared to apo-Lf. In study 2, the investigators want to compare two different dosing regimens, in which they measure iron absorption after one-day washout period and after a two-day washout period, and hypothesize that absorption will be higher after 2 days of washout.

The data from this project will provide valuable information towards the development of new, highly bioavailable iron formulations and dosing regimen that is most efficient.

ELIGIBILITY:
Inclusion Criteria:

* Age of 3-14 months at baseline
* Complementary feeding of the infant has already started
* Assessment of good health as assessed by professional staff at Msambweni District Hospital
* The caregiver is willing to participate in the study
* The informed consent form has been read and signed by the caregiver (or has been read out to the caregiver in case of illiteracy)
* Willingness of the caregiver to provide five blood samples from their child in total during the studies during the visits at the hospital
* Residence in the study for the period of the study

Exclusion Criteria:

* Hb <70 g/L
* Severe underweight (waz <-3)
* Severe wasting (whz <-3)
* Chronic or acute illness or other conditions that in the opinion of the principle investigator or co-researchers would jeopardize the safety or rights of a participant in the trial or would render the participant unable to comply with the protocol
* Participants taking part in other studies requiring the drawing of blood
* Regular intake (>2 days) of iron-containing mineral and vitamin supplements or fortified foods within the last 2 months

Ages: 3 Months to 14 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 25 (Actual)
Dates: Start 2018-12-11 (Actual); Primary Completion 2019-03-30 (Actual); Study Completion 2019-03-30 (Actual)

PRIMARY OUTCOMES:
Fractional iron absorption (%) | Day 21
  Fractional iron absorption from 3 different test meals (apo-, holo-Lactoferrin and FeSO4) erythrocyte incorporation of stable iron isotopes into red blood cells 14 days after test meal

SECONDARY OUTCOMES:
Fractional iron absorption (%) | Day 41
  Fractional iron absorption after 2 different washout periods after receiving test meals (1 day vs 2 days)
Hemoglobin in g/dL (in blood) | Baseline, Day 21, Day 24 (after 1 day washout), Day 27 (after 2 days washout), Day 41
  to identify anemia
Plasma ferritin in µg/L (in blood) | Baseline, Day 21, Day 24 (after 1 day washout), Day 27 (after 2 days washout), Day 41
  to identify iron deficiency
Soluble transferrin receptor in mg/L (in blood) | Baseline, Day 21, Day 24 (after 1 day washout), Day 27 (after 2 days washout), Day 41
  to identify iron deficiency
C-reactive protein in mg/L (in blood) | Baseline, Day 21, Day 24 (after 1 day washout), Day 27 (after 2 days washout), Day 41
  to identify acute inflammation, which inhibits iron absorption
alpha-1-glycoprotein in g/L (in blood) | Baseline, Day 21, Day 24 (after 1 day washout), Day 27 (after 2 days washout), Day 41
  to identify chronic inflammation, which inhibits iron absorption
Plasma hepcidin (in blood) | Baseline, Day 21, Day 24 (after 1 day washout), Day 27 (after 2 days washout), Day 41
  one of major iron absorption regulators

CONTACTS AND LOCATIONS:
Locations (1):
- Msambweni County Referral Hospital, Msambweni, Kwale County, Kenya

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Mikulic N, Uyoga MA, Mwasi E, Stoffel NU, Zeder C, Karanja S, Zimmermann MB. Iron Absorption is Greater from Apo-Lactoferrin and is Similar Between Holo-Lactoferrin and Ferrous Sulfate: Stable Iron Isotope Studies in Kenyan Infants. J Nutr. 2020 Dec 10;150(12):3200-3207. doi: 10.1093/jn/nxaa226. PMID 32886113
- [Derived] Uyoga MA, Mikulic N, Paganini D, Mwasi E, Stoffel NU, Zeder C, Karanja S, Zimmermann MB. The effect of iron dosing schedules on plasma hepcidin and iron absorption in Kenyan infants. Am J Clin Nutr. 2020 Oct 1;112(4):1132-1141. doi: 10.1093/ajcn/nqaa174. PMID 32678434